CLINICAL TRIAL: NCT05892874
Title: Impact of Postoperative Medical Equipment Removal/insertion on Parental Anxiety in Pediatric Cardiac Intensive Care Unit
Status: Completed | Type: Observational
Sponsor: Claude Bernard University (Other)
Collaborators: Research on Healthcare Performance Lab U1290 (Other)
Responsible Party: Principal Investigator, Lilot Marc, Director of research, Claude Bernard University
Other Study IDs: PARANX
Record Dates: First submitted 2023-05-27; First posted 2023-06-07 (Actual); Last update posted 2025-01-28 (Actual); Status verified 2025-01

CONDITIONS: Parents; Anxiety Postoperative

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Month
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Parents

SUMMARY:
A lot of observationnal studies describe parental stressors in PICU/PCICU, but none studied, prospectively, the links between medical equipment removal/insertion and anxiety modulation.

The primary objective is to identify the impact of medical equipment removal/insertion on the STAI-Y score (anxiety) The secondary objective is to identify the parental anxiety determinant (via VAS).

DETAILED DESCRIPTION:
A lot of observationnal studies describe parental stressors in Paediatric Intensive care Unit, but none studied, prospectively, the links between medical equipment removal or insertion and anxiety modulation.

The primary objective is to identify the impact of medical equipment removal or insertion on the STAI-Y score (anxiety) The secondary objective is to identify the parental anxiety determinant (via Visual Analog Stress Scale.

Parents will fill out questionnaire upon arrival in the Intensive care unit when reaching the bedside of their hospitalized child right after the elective cardiac surgery. Then after each equipment removal or insertion they will be asked to fill out again the same questionaire.

ELIGIBILITY:
Inclusion Criteria:

* parents/legal tutor of minor patient (congenital cardiopathy) with elective hospitalization in PCICU for surgical procedures

Exclusion Criteria:

* Parents no french speaking
* child hospitalized for Cardiac Catheterization
* child hospitalized for Berlin Heart insertion
* child hospitalized for heart transplantation

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Parents of minor patients suffering from congenital cardiopathy, hospitalized for electuve surgical procedures
Sampling Method: Non-Probability Sample
Enrollment: 70 (Actual)
Dates: Start 2023-01-30 (Actual); Primary Completion 2024-05-30 (Actual); Study Completion 2024-06-14 (Actual)

PRIMARY OUTCOMES:
State Trait Anxiety Index - Y version | at the arrival in the intensive care unit
  Anxiety declarative scale from 20 to 80 maximum and higher anxiety

SECONDARY OUTCOMES:
Visual Analogic Scale | at the arrival in the intensive care unit
  VAS from 0 to a maximum of 100 mm evaluating: their child confort ; the clinical information's clarity ; their possibility to participate to the care ; the impact on their parental role perceptions ; their trust in caregivers ; their satisfaction concernaing the caregivers attention ; their child clinical condition impacting their (and caregivers) presence in child hospitalization room.

CONTACTS AND LOCATIONS:
Overall Officials: Vincent Piriou, PhD, Study Chair — Hospices Civils of Lyon
Locations (1):
- Unit 11 Hospices Civils of Lyon, Bron, Auvergne-Rhône-Alpes, France

IPD SHARING:
Plan to Share IPD: No